CLINICAL TRIAL: NCT01214096
Title: A Multi-center, Randomized, Double-blind , Placebo Parallel Controlled, Standard Therapy Based Phase III Clinical Trial to Evaluate the Efficacy and Safety of Recombinant Human Neuregulin-1 for Subcutaneous Administration in Patients With Chronic Systolic Heart Failure
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Recombinant Human Neuregulin-1 for Subcutaneous Administration in Patients With Chronic Systolic Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The same protocol has been launched in United States.
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-01-302
Record Dates: First submitted 2010-09-28; First posted 2010-10-04 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart failure; rhNRG-1; MRI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- rhNRG-1 (Experimental): recombinant human neuregulin-1
  Interventions: Drug: rhNRG-1

INTERVENTIONS:
Drug: rhNRG-1 — Subcutaneous Administration:0.6ug/kg/day for 10days
  Arms: rhNRG-1
Drug: rhNRG-1 — Subcutaneous Administration 1.2ug/kg/day for 10 days
  Arms: rhNRG-1
Drug: rhNRG-1 — Vein infusion:0.6ug/kg/day for 10 days
  Arms: rhNRG-1
Drug: placebo — Subcutaneous Administration:0.6 or 1.2ug/kg/day for 10days
  Arms: placebo

SUMMARY:
Evaluate the Efficacy and Safety of Recombinant Human Neuregulin-1 for Subcutaneous Administration in Patients With Chronic Systolic Heart Failure

DETAILED DESCRIPTION:
1. Subcutaneous Administration of NRG-1 is well tolerated by CHF patients
2. Subcutaneous Administration of NRG-1 improves the cardiac function of CHF patients
3. Assessment of relative bioavailability of NRG-1 by Subcutaneous Administration

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, no limitation in gender;
2. Left ventricular ejection fraction (LVEF) ≤ 40% (ECHO);
3. Patients with chronic heart failure (NYHA class II or III);
4. In the past one month, the clinical condition (including history, clinical symptoms and signs) was relatively stable;
5. Patients on standard treatment of chronic heart failure at the target dose or maximum tolerance dose for over 1 month ,or unchanged dose in last 1 month;
6. Understand and sign the informed consent form;

Exclusion Criteria:

1. Atrial fibrillation;
2. Subject underwent cardiac pacemaker treatment;
3. Subject underwent metal graft treatment;
4. Claustrophobia;
5. Acute myocardial infarction, cardiac ischemia indicated by 6-minute walk test, hypertrophic cardiomyopathy, constrictive pericarditis, significant valve disease or congenital heart disease, severe pulmonary hypertension;
6. Ischemic heart failure without the revascularization or undergone the revascularization within last 6 months;
7. Subject underwent cardiac surgery or cerebrovascular events within the previous six months;
8. Subjects who plan to have cardiac transplantation;
9. Severe hepatic and renal insufficiency (serum creatinine>2.0 mg /dl, AST or ALT is five times higher than the upper limit of normal range);
10. Subject needs mechanical ventilation;
11. Systolic blood pressure < 90mmHg, or > 160mmHg;
12. Chronic heart failure complicated with acute hemodynamic disturbance or acute decompensation within last 1 month;
13. Mobitz Type II or III° atrial ventricular block，severe ventricular arrhythmia (polymorphic and frequent premature ventricular beats, frequent non-sustained ventricular tachycardia);
14. Serum potassium<3.2mmol/L, or>5.5mmol/L;
15. Female subject is pregnant or plan to become pregnant
16. Childbearing-aged female subject who is unmarried or dose not bear child;
17. Subject with life expectancy less than 6 months as assessed by investigators;
18. Subject participated in any other clinical trial within the previous three months;
19. Subject with previous history of tumor, or current tumor patient, or subject with pre-cancerous disease manifested by pathological examination (such as ductal carcinoma in situ or cervical epithelial dysplasia)
20. Examinations (physical examination, X-ray examination, type-B ultrasonic detection or other methods) reveal that the subject has malignant mass, gland hyperplasia or adenoma with endocrine activity, or impact on heart, or endocrine function (such as pheochromocytoma, thyroid enlargement);
21. The Investigator deemed for whatever reason that the subject is not likely to complete the study or comply with the study procedures (due to administration or any other reason).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
cardiac function measured by MRI | 30 days

SECONDARY OUTCOMES:
cardiac function | baseline, 30 days, 90day and180 days
  6-minute walk test, cardiac function classification(NYHA)，life quality score.

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Principal Investigator — Cardiovascular Institute and Fuwai Hospital
Locations (4):
- China (4):
  - Beijing Anzhen Hospital of Capital University of Medical Sciences, Beijing
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Cardiovascular Institute & Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - General Hospital of People's Liberation Army, Beijing